CLINICAL TRIAL: NCT06159907
Title: Evaluation of the Diagnostic and Prognostic Role of PET (PET/CT and PET/MRI) in Gynecological Tumors.
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PET-GYN-Retrospective
Record Dates: First submitted 2023-11-27; First posted 2023-12-07 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Gynecological Tumors
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: the diagnostic and prognostic value of PET/MRI and PET/CT with 18F-FDG in patients presenting with gynecological tumors — For the evaluation of patients affected by endometrial cancer, the correlations between semi-quantitative PET parameters (SUVmax, SUVmean, MTV and TLG calculated at different SUVmax thresholds) and histological data, such as for example myometrial invasion, will be investigated. lymph node invasion, tumor grade and type, risk level, probability of mutation of the p53 gene, etc.
  In addition to traditional imaging parameters we will also investigate the usefulness of radiomic features, i.e. quantitative data extracted from PET images (PET/CT or PET/MRI), in predicting and explaining histological data

SUMMARY:
Gynecological cancers involve several tumors of the female reproductive system. The five most common gynecological tumors are those of the uterine cervix, endometrium, ovary, vagina and vulva. Furthermore, although rarer, there is a further gynecological tumor, which is generated from the gestational trophoblast tissue.These pathologies represent an important burden for society since there are over nine hundred thousand cases in Europe.

Ultrasound examination is the investigation commonly used to monitor high-risk women.

Magnetic resonance imaging (MRI) is considered the most accurate imaging technique for presurgical staging of gynecological tumors. Computed tomography (CT), on the other hand, is not usually used for diagnosis, but is considered very useful for investigating possible distant metastases.Finally, integrated positron emission tomography (PET)/CT and PET/MRI methods are innovative molecular imaging techniques and represent a continually expanding field of research in the oncology setting, including gynecological malignancies.

The present study is of considerable clinical relevance as at our Institute it is possible to have a significant number of patients suffering from gynecological neoplastic pathologies that are studied using PET, thus allowing the identification and validation of innovative imaging biomarkers, with the use of both traditional imaging parameters and radiomic features.

ELIGIBILITY:
Inclusion Criteria:

* adult patients suffering from a gynecological oncological disease; Patients who have performed at least one PET study with 18F FDG for the staging or restaging of their oncological pathology; patients who give written informed consent to the study

Exclusion Criteria:

* patients <18 years lack of availability of clinical and PET imaging data useful for analyses.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: In this study, all patients referred to the gynecology oncology unit of the IRCCS San Raffaele from 01/01/2009 to July 2021 who underwent a PET examination with 18 F FDG at the unit of Nuclear Medicine at the IRCCS San Raffaele for clinical reasons will be considered.
Sampling Method: Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2024-12-27 (Estimated); Study Completion 2024-12-27 (Estimated)

PRIMARY OUTCOMES:
PET/MRI and PET/CT with 18F-FDG in patients with gynecological tumors. | 3 year
  Integrated positron emission tomography (PET)/CT and PET/MRI methods are innovative molecular imaging techniques are able to provide information in predicting and explaining histological data in gynecological tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: No